CLINICAL TRIAL: NCT02898493
Title: Translation, Cultural Adaptation and Validation of the Creole Versions of the EQ-5D and the SF-36 Questionnaires in Patients With Type II Diabetes in Reunion Island, Martinique and Guadeloupe
Acronym: CreoQol
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/CHU/09
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Validation of questionnaire; Quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The evaluation of quality of life in health is particularly important for measuring the impact of the chronic diseases. The scales of measure constitute the main measurement tool in clinical trials because of their psychometrics properties and of their ease of use.

Among these scales, the 36-Item Short Form Survey (SF-36) and the EuroQol five dimensions questionnaire ( EQ-5D) were widely validated in various populations, of which the population of the diabetics patients. Both scales have validated versions in French.

In the Antilles and in Reunion Island, diabetes is a frequent pathology and is the subject of many clinical and epidemiological trials. One of the difficulties encountered during the implementation of these studies is the absence of measurement tools validated for these populations.

Investigators thus suggest, within a common workgroup uniting Guadeloupe, Martinique and Reunion Island, adapting and validating these scales according to an identical procedure in Creole from Guadeloupe, from Martinique and from Reunion Island and validating the French versions of these scales in their populations of type II diabetics patients.

ELIGIBILITY:
Inclusion Criteria:

* male or female ≥ 18 years of age
* type II diabetes diagnosed more than 1 year ago
* creole speaking
* living on the island for more than 5 years
* agreed and signed the informed consent form

Exclusion Criteria:

* not able to understand and follow the instructions
* patients with proven cognitive issues which do not make possible to complete questionnaire
* patients with current acute and serious complications associated with diabetes
* medical history of stroke with physical or neurological damage
* patients already involved in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type II diabetic patients seen in the department of diabetology at the University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Internal Consistency (IC) assessed as Cronbach's Alpha Value | 1 day (inclusion day)

SECONDARY OUTCOMES:
Test-retest Reliability | 3-4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Reunion Island, Saint-Denis, Reunion Island, France